CLINICAL TRIAL: NCT06181019
Title: Acupuncture Combined With Mirabegron in the Treatment of Overactive Bladder Syndrome: A Prospective Randomized Controlled Trial
Brief Title: Acupuncture Combined With Mirabegron in the Treatment of OAB
Acronym: ACWMITTOOAB
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Affiliated Ganzhou Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Huang Xin, Associate Senior Doctor, The Affiliated Ganzhou Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TY-ZKY-2023-045-01
Record Dates: First submitted 2023-12-11; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; mirabegron; acupuncture; nocturia; incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Nocturia | interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: Patients in the control group were treated with 50 mg of mirabegron (Astellas Pharma, Tokyo, Japan) for 12 weeks, whereas patients in the treatment group were treated with acupuncture combined with mirabegron.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Be treated with mirabegron. (Active Comparator): Patients were treated with 50 mg of mirabegron (Astellas Pharma, Tokyo, Japan) for 12 weeks.
  Interventions: Drug: 50 mg of mirabegron
- Be treated with acupuncture combined with mirabegron. (Experimental): Patients were treated with acupuncture combined with mirabegron.
  Interventions: Combination Product: acupuncture combined with mirabegron.

INTERVENTIONS:
Drug: 50 mg of mirabegron — Patients in the control group were treated with 50 mg of mirabegron (Astellas Pharma, Tokyo, Japan) for 12 weeks.
  Other Names: mirabegron
  Arms: Be treated with mirabegron.
Combination Product: acupuncture combined with mirabegron. — Patients in the treatment group were treated with acupuncture combined with mirabegron.
  Arms: Be treated with acupuncture combined with mirabegron.

SUMMARY:
Introduction: As conventional treatments for overactive bladder (OAB) have not yet shown satisfactory results, new approaches are needed. Therefore, this study aimed to investigate the efficacy and safety of acupuncture combined with mirabegron for the treatment of OAB.

Methods: This prospective cohort study enrolled 80 OAB patients who were then divided into control and treatment groups using a randomized number-table method. The control group was administered mirabegron alone (50 mg/day), while the treatment group was administered mirabegron orally along with acupuncture at the following points: guanyuan (CV4), zhongji (CV3), and sanyinjiao (SP6). The OAB symptom score (overactive bladder syndrome score [OABSS]), voiding, urgency, nocturia, incontinence, and incidence of related adverse events were compared between the two groups at baseline and after 4, 8, and 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of OAB
* Good compliance
* Good communication skills

Exclusion Criteria:

* Age <14 or >75 years
* History of use of M-blockers in the recent 4-6 weeks
* History of use of α-blockers in the recent 4-6 weeks
* History of use of mirabegron in the recent 4-6 weeks
* Diagnosis with a combined urinary tract tumor
* Inability to cooperate with this study
* Pregnancy
* Postvoid residual urine volume >150 mL

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overactive bladder syndrome scores (OABSS) | 4, 8, and 12 weeks after treatment
  overactive bladder syndrome scores of patient
voiding diary indicators (voiding, urgency, nocturia, and incontinence) | 4, 8, and 12 weeks after treatment
  Number of voiding, urgency, nocturia, and incontinence in one day

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Deng, M.D., Principal Investigator — Ganzhou People's Hospital
Locations (1):
- Ganzhou People's Hospital, Ganzhou, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided